CLINICAL TRIAL: NCT05892211
Title: The Pilot Study of LINE-1 and Alu Methylation Levels Among Middle Aged Women With Low Cardiovascular Risk Profile in Respect of Menopausal Hot Flashes
Brief Title: LINE-1 and Alu Methylation Levels Among Middle Aged Women With Low Cardiovascular Risk Profile in Respect of Menopausal Hot Flashes
Status: Suspended | Type: Observational
Why Stopped: The university has relocated to a new place due to earthquake.
Sponsor: Istanbul University - Cerrahpasa (Other)
Collaborators: Scientific Research Project Coordination Unit of Istanbul University-Cerrahpasa (Unknown)
Responsible Party: Principal Investigator, Ipek B. Ozcivit Erkan, MD, Resident Doctor, Istanbul University - Cerrahpasa
Other Study IDs: E-83045809-604.01.02-3916
Record Dates: First submitted 2023-05-09; First posted 2023-06-07 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Hot Flashes; Sleep; Menopause; Cardiovascular Diseases; Epigenetics; DNA Methylation
Keywords: DNA methylation; Hot Flashes; Sleep; Vasomotor symptoms; Menopause; Cardiovascular Diseases; epigenetics
MeSH Terms: conditions — Hot Flashes; Cardiovascular Diseases | interventions — Polysomnography; Galvanic Skin Response

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — 2 cc peripherical venous blood specimens were obtained from the participants into EDTA blood collection tubes. DNA was isolated by Nucleospin Blood Kit.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1 (vasomotor symptoms present): Participants who have vasomotor symptoms. Sleep is recorded by polysomnography for a night. Hot flashes during sleep are recorded by two electrodes measuring the skin conductance near sternum. Any hot flashes reported subjectively by the patient during the recording is noted. Their blood samples are obtained.
  Interventions: Diagnostic Test: Polysomnography; Diagnostic Test: Skin conductance; Genetic: ALU and LINE-1 DNA methylation analysis; Diagnostic Test: The Menopause-Specific Quality of Life Questionnaire (MENQOL); Diagnostic Test: Pittsburgh Sleep Quality Index (PSQI)
- Group 2 (vasomotor symptoms absent): Participants who don't have vasomotor symptoms. Sleep is recorded by polysomnography for a night. Hot flashes during sleep are recorded by two electrodes measuring the skin conductance near sternum. Any hot flashes reported subjectively by the patient during the recording is noted. Their blood samples are obtained.
  Interventions: Diagnostic Test: Polysomnography; Diagnostic Test: Skin conductance; Genetic: ALU and LINE-1 DNA methylation analysis; Diagnostic Test: The Menopause-Specific Quality of Life Questionnaire (MENQOL); Diagnostic Test: Pittsburgh Sleep Quality Index (PSQI)

INTERVENTIONS:
Diagnostic Test: Polysomnography — Polysomnography is performed by 3-channel electroencephalography ((EEG; F4-M1, C4-M1, O2-M1), 2-channel electrooculography (EOG), chin electromyography (EMG), surface EMG recording from tibialis anterior muscles of the right and left leg, body position, oronasal thermal airflow sensor, nasal pressure sensor, thoracic and abdominal respiratory belts for assesing the respiratory effort, electrocardiography (ECG), pulse, recording of respiratory sounds, oxygen saturation and synchronous video recording. The sleep stages are scored by the current criteria of American Academy of Sleep Medicine.
Diagnostic Test: Skin conductance — The sympathetic skin response recordings are performed with a four-channel electromyography apparatus (Nihon-Kohden). They are recorded from both sides of the sternum with the active and reference electrodes placed 2 cm apart from the midline.
Genetic: ALU and LINE-1 DNA methylation analysis — 2 cc peripheric venous blood is drawn from the participants to the test tubes with EDTA. DNA isolation is done by Nucleospin Blood Kit (REF:740951.250, Macherey-Nagel). Epitect Fast DNA Bisulfite Kit (REF:59824, Qiagen) is used to do DNA bisulfite modification. ALU and LINE-1 site specific methylation primer is designed and the methylation patterns are compared between the groups by Epitect Methylight PCR Kit (Cat. No:59496, Qiagen).
Diagnostic Test: The Menopause-Specific Quality of Life Questionnaire (MENQOL) — The Menopause-Specific Quality of Life Questionnaire (MENQOL) is filled by each participant to assess the health related quality of life before the polysomnography test.
Diagnostic Test: Pittsburgh Sleep Quality Index (PSQI) — Pittsburgh Sleep Quality Index (PSQI) is done by each participant to assess the sleep quality and disturbances before thepolysomnography test.

SUMMARY:
Vasomotor symptoms are the most common symptoms seen during climacterium. The hypoestrogenic state causes dysfunction of hypothalamic preoptic area, a thermoregulatory center. The sympathetic overactivation during the hot flashes is associated with awakening during sleep and have a negative impact on cardiac indexes and vascular reactivity. Therefore, hot flashes are accepted as subclinical cardiovascular risk factor.

The association between the severity of the hot flashes and cardiovascular risk may have an epigenetic background. Recently, methylation changes of DNA was found to be associated with clinical and subclinical cardiovascular disease risk (atherosclerosis and hypertension etc.). A transposable element in the DNA, Long interspersed nuclear elements (LINE-1), was found to be hypomethylated in cases with ischemic heart disease and stroke. Therefore, the expression of repeating elements in the DNA (LINE-1 and ALU) may be considered as a mediator in the ischemic heart disease. Until now, menopausal age, vasomotor symptoms and epigenetic and biological aging have been evaluated. However, the epigenetic impact of severe vasomotor symptoms in postmenopausal women with low cardiovascular disease risk profile has not been evaluated. In this study, we aimed to evaluate the epigenetic basis of cardiovascular disease risk for women with vasomotor symptoms which disturb sleep by assessing the methylation levels of ALU and LINE-1.

DETAILED DESCRIPTION:
Vasomotor symptoms are the most common symptoms seen during climacterium. The hypoestrogenic state causes dysfunction of hypothalamic preoptic area, a thermoregulatory center. The variations in the range of thermoneutral zone determine the severity of the vasomotor symptoms. Sympathetic overactivation during the hot flash and decreased rate of parasympathetic control on the heart rate are the main factors contributing to the cardiovascular disease risk. The hot flashes which occur and cause awakening during sleep have negative impact on cardiac indexes and vascular reactivity. Therefore, vasomotor symptoms are accepted as subclinical cardiovascular risk factor.

Hot flashes associated with nighttime awakenings were shown to increase systolic and diastolic blood pressure and decrease pre-ejection period. Objectively recorded hot flashes and nighttime awakenings were found to be correlated white matter hyperintensities in the brain which show poor brain health. In addition, white matter hyperintensities may be considered as a cerebral small vascular disease and is associated with greater odds of having stroke and dementia.

Among postmenopausal women, cardiovascular disease is the most prevalent cause for mortality and morbidity. It results from the interaction of environmental and genetic factors. The association between the severity of hot flashes and cardiovascular risk may have an epigenetic background. The global DNA methylations were found to be decreased in postmenopausal women with high cardiovascular disease risk. Recently, methylation changes of DNA was found to be associated with clinical and subclinical cardiovascular disease risk (atherosclerosis and hypertension etc.). A transposable element in the DNA, Long interspersed nuclear elements (LINE-1), was found to be hypomethylated in cases with ischemic heart disease and stroke. Therefore, the expression of repeating elements in the DNA (LINE-1 and ALU) may be considered a mediator in the ischemic heart disease. Until now, menopausal age, vasomotor symptoms and epigenetic and biological aging have been evaluated. However, the epigenetic impact of severe vasomotor symptoms in postmenopausal women with low cardiovascular disease risk profile has not been evaluated. In this study, we aimed to evaluate the epigenetic basis of cardiovascular disease risk for women who have low cardiovascular disease risk profile at baseline and have vasomotor symptoms which disturb sleep by assessing the methylation levels of ALU and LINE-1.

ELIGIBILITY:
Inclusion Criteria:

* 45-55 years of age
* Women with serum FSH levels >35 IU/L, serum estradiol levels <20 pg/mL
* Women with low cardiovascular disease risk profile (Framingham score for coronary heart disease <10%),
* Low high sensitive CRP levels (<5 mg/L),
* Fasting glucose <90 mg/dL,
* Fasting levels of insulin <37.06 µIU/mL,
* Blood pressure <140/90 mmHg (measured 2 times with 10 minutes interval),
* TSH <4.2 mIU/L and fT4 <1.7 ng/dL,
* Hemoglobin levels 12-16 g/dL, leucocyte count <10.3*10^3/µL and neutrophil count <4.9*10^3/µL; eosinophil count <0.5*10^3/µL, basophil count <0.2*10^3/µL

Exclusion Criteria:

* Women with high cardiovascular disease risk profile (Framingham score for coronary heart disease >10%),
* Women who were diagnosed with a cardiovascular disease (coronary heart disease, stroke),
* Women with hypertension,
* Smokers,
* BMI >30 kg/m2,
* Women with diabetes
* Women who were surgically postmenopausal,
* Women who used hormone therapy in the last three months,
* Women with obstructive sleep apnea
* Women who are using medicine which may cause sleep disturbances.

Ages: 45 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study population consists of women aged between 45-55 with low cardiovascular disease risk profile assessed by Framingham score system. The study population doesn't include any women who were already diagnosed with hypertension, coronary heart disease, diabetes, obstructive sleep apnea and stroke. It is a very homogenous population in terms of baseline cardiovascular disease risk apart from the presence or absence of hot flashes.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2032-03-08 (Estimated)

PRIMARY OUTCOMES:
Methylation levels of ALU and LINE-1 | 1 day
  Methylation levels of ALU and LINE-1 in women with vasomotor symptoms
Polysomnographic findings | 1 night
  Total sleep time in women with vasomotor symptoms
Number of objective hot flashes per night | 1 night
  Number of objective hot flashes per night measured by sternal skin conductance in women with vasomotor symptoms
Number of nighttime awakenings per night | 1 night
  Number of nighttime awakenings per night associated with hot flash episodes
Polysomnographic findings | 1 night
  Sleep efficiency in women with vasomotor symptoms
Polysomnographic findings | 1 night
  Sleep stages in women with vasomotor symptoms

SECONDARY OUTCOMES:
Subjective sleep findings (Pittsburgh Sleep Quality Index (PSQI)) | 1 night
  Scores of PSQI questionnaire in women with vasomotor symptoms (>5 can be considered as a significant sleep disturbance.)
Menopause-Specific Quality of Life Questionnaire (MENQOL) scores and its association with hot flashes per night | 1 day
  Scores of MENQOL and its association with hot flashes per night (There is no limit, higher scores on the MENQOL indicate a poorer quality of life.)

CONTACTS AND LOCATIONS:
Overall Officials: Ipek Betul Ozcivit Erkan, MD, Principal Investigator — Istanbul University - Cerrahpasa
Locations (1):
- Istanbul University-Cerrahpasa, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
The data could be shared on demand.